CLINICAL TRIAL: NCT07167992
Title: Comparison of Talc Slurry Versus Talc Insufflation: A Study on Effectiveness, Safety, and Hospital Outcomes in Pleurodesis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Zeeshan Sarwar, Principal Investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB/2025/1559/SIMS
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Pneumothorax Spontaneous Primary; Pneumothorax Spontaneous Secondary; Pleural Effusion, Malignant; Pleurodesis
Keywords: Talc slurry; Talc Insufflation; Pleurodesis; malignant pleural effusions; recurrent pneumothorax
MeSH Terms: conditions — Pneumothorax; Pleural Effusion, Malignant | interventions — Pleurodesis

STUDY DESIGN:
Intervention Model Description: This study will be a randomized controlled trial (RCT) to ensure robust comparisons between talc slurry (TS) and talc insufflation (TI) in managing pleural effusions or pneumothoraces. To reduce bias, the study will be single-blind, where patients will be unaware of the procedure type, while clinicians will know the intervention. This design minimizes performance and response biases without compromising the feasibility of the procedures.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Talc Slurry Group (Experimental): patient undergoing pleurodesis by talc slurry method are included in this group
  Interventions: Procedure: Pleurodesis
- Talc Insufflation Group (Experimental): patient undergoing pleurodesis by talc insufflation method are included in this group
  Interventions: Procedure: pleurodesis

INTERVENTIONS:
Procedure: Pleurodesis — Talc slurry pleurodesis is a chemical technique for managing recurrent pleural effusions and pneumothoraces. The procedure involves instilling a suspension of talc (4-5 grams) in sterile saline (50-100 mL) into the pleural space via a chest tube. This induces an inflammatory reaction, leading to fibrosis and fusion of pleural surfaces. The technique demonstrates 70-90% success rates in malignant pleural effusions and pneumothoraces, with efficacy comparable to talc poudrage. While generally safe, potential complications include pain, fever, and rarely, pneumonitis or empyema. Use of large-particle, asbestos-free talc and standardized protocols has improved its safety profile.
  Arms: Talc Slurry Group
Procedure: pleurodesis — Talc insufflation, is a pleurodesis technique involving direct insufflation of dry talc powder into the pleural cavity during thoracoscopy. It allows visual inspection of the pleural space and concurrent diagnostic procedures. Success rates range from 85% to 93% for malignant pleural effusions and pneumothoraces, with efficacy comparable or potentially superior to talc slurry in some studies. The procedure typically requires general anesthesia and is more invasive than talc slurry. Common side effects include chest pain, fever, and dyspnea. The risk of severe respiratory complications has decreased with large-particle, asbestos-free talc. While effective, the choice between insufflation and slurry depends on patient factors, institutional expertise, and resource availability.
  Arms: Talc Insufflation Group

SUMMARY:
Pleural effusion is characterized by the accumulation of fluid in the pleural space, which typically contains about 10-20 mL of pleural fluid that is crucial for the movement of the lungs against the chest wall. This fluid closely resembles plasma but has a lower protein concentration, usually less than 1.5 gm/dL. It primarily originates from pleural capillaries and the interstitial spaces of the lung, and is reabsorbed through the lymphatic vessels in the parietal pleura, either via small openings known as stomas or through a process called transcytosis (1, 2). When the balance between fluid production and reabsorption is disrupted-often due to various pathogenic mechanisms-it can lead to pleural effusion. In such cases, effective management is essential. This study aims to conduct a thorough comparison of the two talc administration methods-TS and TI-using sterilized, large-particle, asbestos-free talc powder. By examining key outcome measures such as pleurodesis success rates, procedural morbidity, and length of hospital stay, the goal is to provide clinicians with evidence-based guidance to facilitate informed decision-making in the management of pleural effusions.

DETAILED DESCRIPTION:
One of the most effective interventions for managing malignant pleural effusion (MPE) and pneumothoraces is chemical pleurodesis, which involves the introduction of a sclerosing agent into the pleural space to induce inflammation and subsequent fibrosis, thereby closing the pleural space. Among the various agents used, talc is the most widely recognized for its high success rates, affordability, and availability (3-8). There are primarily two methods of delivering talc: talc slurry (TS), which involves injecting a talc suspension via a chest tube, and talc insufflation (TI), which is performed during thoracoscopic surgery. Currently, there is no consensus on which method is superior, leading to a recommendation for individualized patient approaches that consider the specific clinical scenario and aim to minimize complications while reducing hospital stays9 .

The choice of talc particle size is critical, as it has significant implications for both the efficacy of pleurodesis and the safety of the procedure. Historically, small-particle talc formulations (less than 10 μm) have been associated with severe complications such as acute respiratory distress syndrome (ARDS) 10. This has prompted a shift toward using larger particles (greater than 15 μm), which have been shown to decrease the risk of ARDS and other respiratory complications. Importantly, studies have demonstrated that the effectiveness of pleurodesis is not compromised by the use of larger particles11.Furthermore, recommendations now advocate for the use of a minimum effective dose of talc, typically around 4-5 grams, to optimize both efficacy and safety.

Another significant advancement in the use of talc for pleurodesis is the transition to asbestos-free formulations. Historically, some talc preparations contained trace amounts of asbestos, a known carcinogen linked to serious health risks such as mesothelioma. The move toward asbestos-free talc has been driven by the need to eliminate these long-term carcinogenic risks, especially in patients who may have a prolonged survival following pleurodesis. Despite significant advancements in the use of talc pleurodesis, several important gaps remain in the literature. Notably, there is a lack of comprehensive studies focusing on the efficacy and safety of large-particle (≥15 μm), asbestos-free talc. While this formulation has been associated with a reduced risk of complications such as acute respiratory distress syndrome (ARDS), most existing research has centered on smaller-particle talc or formulations with less stringent quality controls. Furthermore, the comparative effectiveness of talc slurry (TS) and talc insufflation (TI) using modern, large-particle, asbestos-free talc is underexplored. The absence of such data hinders the development of evidence-based guidelines for selecting the optimal delivery method for individual clinical scenarios While these advancements have improved the risk-benefit profile of talc pleurodesis, it is important to recognize that the procedure is not without risks. Thus, careful patient selection and monitoring remain essential to minimize complications 12. Reducing hospital stays and procedural morbidity is critical in improving patient outcomes, especially for individuals with malignant pleural effusion (MPE) or recurrent pneumothoraces. These conditions often affect patients with advanced malignancies or significant comorbidities, where maintaining quality of life is paramount. Shorter hospital stays and fewer complications directly enhance patients' overall well-being and comfort, particularly for those with limited life expectancy. Additionally, minimizing hospital stays alleviates the economic and logistical burdens on healthcare systems, promoting the broader implementation of pleurodesis as a sustainable intervention.

International guidelines, such as those issued by the British Thoracic Society (BTS), provide valuable insights into the current standards of care for pleurodesis. These guidelines recommend talc pleurodesis as a primary intervention for symptomatic management of recurrent pleural effusions and pneumothoraces when pleural drainage alone proves insufficient. Talc remains the preferred agent due to its high efficacy and relative safety profile. However, the BTS guidelines do not strongly favor one delivery method-talc slurry or talc insufflation-over the other, advocating instead for individualized approaches based on patient needs and resource availability. The guidelines emphasize the importance of using sterilized, asbestos-free, large-particle talc to reduce the risk of complications, including ARDS and long-term carcinogenic effects13.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 12 years and older.
* Diagnosed with malignant pleural effusions or pneumothoraces.
* ECOG performance status of 0-2.
* Life expectancy of at least 3 months.
* Ability to provide informed consent.
* No contraindications to general anesthesia or conscious sedation.

Exclusion Criteria:

* Patients younger than 12 years old
* Female patients who are pregnant or lactating
* Patients with encysted or septated pleural effusions and pneumothoraces
* Patients presenting with respiratory failure
* Patients complaining of dyspnea in spite of complete evacuation of pleural effusion or pneumothorax.
* Patients with evident chest infection with clinical or laboratory signs suggestive of parapneumonic effusions.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Success of Pleurodesis | 01 months post-procedure
  The success rate of pleurodesis is defined as the percentage of patients who achieve complete resolution of pleural effusion or pneumothorax within a specified time frame of 01 months post-procedure. Success is assessed through follow-up chest radiographs, with criteria for success including the absence of fluid reaccumulation or lung collapse during this period. Clinical improvement in symptoms such as dyspnea may also be considered as supplementary evidence of a successful outcome.

SECONDARY OUTCOMES:
Procedural Morbidity of pleurodesis | 30 days
  Procedural morbidity refers to the incidence and severity of complications directly attributable to the pleurodesis procedure, occurring within 30 days post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Shoaib Nabi, Professor of Thoracic Surgery, Study Chair — Services institute of Medical Sciences (SIMS), Services Hospital Lahore
Locations (1):
- Services Institute of Medical Sciences (SIMS), Services Hospital Lahore, Lahore, Punjab Province, Pakistan